CLINICAL TRIAL: NCT04000490
Title: Validation of the SCARE Score, Predictive Score of Acute Coronary Syndrome During the Assessment of Chest Pain in the Call Center.
Brief Title: External Validation of the SCARE Score
Acronym: SCARE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: CHRO-2019-05
Record Dates: First submitted 2019-06-07; First posted 2019-06-27 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Assessment; Chest Pain; ACS - Acute Coronary Syndrome
Keywords: Assessment; chest pain; ACS predictive score; physician's belief
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with a chest pain: adult patient with a chest pain calling for urgency center
  Interventions: Other: SCARE Score

INTERVENTIONS:
Other: SCARE Score — Predictive Score of acute coronary syndrome during the medical assessment of chest pain

SUMMARY:
Chest pain is a very common reason for resorting to the call center. The etiologies are very varied, ranging from benign pathologies to some that may involve, in the short term, the vital prognosis such as Acute Coronary Syndrome (ACS). ACS is a partial or complete occlusion of a coronary artery that causes potentially irreversible myocardial pain unless prompt treatment is undertaken. ACS represents 120 000 cases per year in France and causes about 18 000 deaths. There is currently no support score for the assessment of chest pain. However, reducing the duration of management of ACS is essential in order to hope to reduce the associated morbidity and mortality. In 2016, SAMU45's team established a predictive ACS score for the assessement of chest pain in SAMU 45 (France) based on the prospective study of 1367 patients. Seven items significantly associated with this risk of ACS could be highlighted: age, sex, smoking, typicality (potentially constrictive chest pain radiating potentially to the shoulders and / or jaw) pain, inaugural character of pain (ie first episode of this type), presence of sweats and the physician's belief to be in the presence of an ACS. These seven variables make up the SCARE score. This had good internal discrimination (AUC at 0.81) and excellent calibration ("p" of Hosmer-Lemeshow at 0.74). This score makes it possible to stratify the risk of ACS, by using epidemiological elements but also the physician's belief, whose Negative Predictive Value (VPN) proved excellent.

The objective of this new project is to confirm by an external validation via a multicentric study the robustness of this score and thus be able to consider its use in front of any chest pain regulated in France by a call center.

DETAILED DESCRIPTION:
The main objective is to validate the predictive SCARE score of acute coronary syndrome during the medical assessment of chest pain. The primary endpoint will be SCARE score analysis (pre-established in 2016) with assessment of its calibration (Hosmer Lemeshow) and discrimination (AUC) in a multicenter population of chest pain with a potential diagnosis of Acute Coronary Syndrome established according to the European Society of Cardiology criteria.

This is a multi-center study including any patient over 18 years of age calling call center for chest pain over a period of six months. It will exclude post-traumatic chest pain, patients under 18 years old, patients who do not speak French, patients refusing to participate in the study or refusing treatment, patients not affiliated to social security, patients incarcerated in a penitentiary center, patients under tutorship, curatorship or safeguard of justice.

The collection of data will be carried out thanks to files filled prospectively by the medical physician for each call for the reason of a chest pain. These cards will list the epidemiological data (age, sex, weight, height) and clinical data of each patient, as well as the decision and the resources committed by the regulating physician (hospital care via SMUR or ambulance, treatment in city medicine). For hospitalized patients, the diagnosis of ACS will be retained if the patient meets the criteria defined by the European Society of Cardiology. For patients managed in ambulatory medicine, a telephone call to the patient will be made at one month to obtain the diagnosis.

Then, the SCARE score will be analized in this multicenter population with evaluation of its calibration (Hosmer Lemeshow) and discrimination (AUC). The characteristic performances of the score (sensitivity, specificity, PPV, NPV, positive and negative likelihood ratios)will also be analized.

ELIGIBILITY:
Inclusion Criteria:

* Any patient over the age of 18 calling call center for chest pain

No-inclusion Criteria:

* Posttraumatic chest pain,
* Age under 18,
* Patient not speaking French,
* Patient refusing to participate in the study or refusing care
* Patient not affiliated with social security,
* Patients incarcerated in a penitentiary center,
* Patients under guardianship, curatorship or safeguard of justice.

Exclusion Criteria:

- Patient refusing to participate in the study or refusing care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient over the age of 18 calling call center for chest pain
Sampling Method: Non-Probability Sample
Enrollment: 2205 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
SCARE score with evaluation of its calibration and its discrimination in a multicentric population | up to one month
  Data will be collected during each patient's call for chest pain. Epidemilogical data (age, sex, weight, height) and clinical data will be collected, as well as the decision and the ressources committed by the regulating physician. For hospitalized patients, the diagnosis of acute coronary sydrom will be retained if patient meets the criteria defined by the European Society of Cardiology. For patients managed in ambulatory médicine, a telephone call to the patient will be made at one month in order to obtain the diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey GUERINEAU, MD, Principal Investigator — CHR Orléans; Paul Louis MARTIN, MD, Principal Investigator — CHRU Tours - hopital trousseau; Thomas MOUMNEH, MD, Principal Investigator — University Hospital, Angers; Jeremy GUENEZAN, MD, Principal Investigator — CHU Poitiers
Locations (4):
- France (4):
  - CHU Angers, Angers
  - CHRU de Tours, Chambray-lès-Tours
  - CHR d'Orléans, Orléans
  - CHU poitiers, Poitiers

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faxon D, Lenfant C. Timing is everything: motivating patients to call 9-1-1 at onset of acute myocardial infarction. Circulation. 2001 Sep 11;104(11):1210-1. No abstract available. PMID 11551867
- [Background] Mathew TP, Menown IB, McCarty D, Gracey H, Hill L, Adgey AA. Impact of pre-hospital care in patients with acute myocardial infarction compared with those first managed in-hospital. Eur Heart J. 2003 Jan;24(2):161-71. doi: 10.1016/s0195-668x(02)00521-3. PMID 12573273
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Katus HA, Lindahl B, Morrow DA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S. Third universal definition of myocardial infarction. Circulation. 2012 Oct 16;126(16):2020-35. doi: 10.1161/CIR.0b013e31826e1058. Epub 2012 Aug 24. No abstract available. PMID 22923432
- See also: thesis : Syndrome Coronarien Aigu (SCA) lors de la REgulation d'un appel au Centre 15 pour douleur thoracique : le score SCARE — http://memoires.scd.univ-tours.fr/Medecine/Theses/2017_Medecine_GuerineauAudrey.pdf